CLINICAL TRIAL: NCT05001997
Title: Effects of Lactose-free Dairy Products on Athletes With Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Central Lancashire (Other)
Responsible Party: Principal Investigator, Jan Mei Soon, Senior Lecturer, University of Central Lancashire
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HEALTH 0158
Record Dates: First submitted 2021-07-26; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Single-blinded, randomised crossover study
Who Masked: Participant
Masking Description: All yogurt labels will be covered or masked with corrugated sleeves
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet A - Lactose free probiotic yogurt (Active Comparator): Plain flavoured lactose free probiotic yogurt (contains Lactobacillus acidophilus and Bifidobacterium lactis)
  Interventions: Dietary Supplement: Lactose free probiotic yogurt
- Diet B - Lactose free yogurt (non-probiotic) (Placebo Comparator): Plain flavoured lactose free yogurt (contains only starter cultures)
  Interventions: Dietary Supplement: Lactose free probiotic yogurt

INTERVENTIONS:
Dietary Supplement: Lactose free probiotic yogurt — Probiotics are non-pathogenic, live microbes that when eaten or administered In adequate amount, it confer health benefits to host. Only lactose free probiotic yogurt containing cultures such as Lactobacillus acidophilus and Bifidobacterium lactis will be selected.

SUMMARY:
Irritable Bowel Syndrome (IBS) is a gastrointestinal disorder defined by recurrent abdominal pain, bloating, abdominal distention and altered bowel habits. IBS is common among athletes and can impair performance. IBS was found to be prevalent in 9.8% (n=430) of endurance athletes. The condition is associated with significantly reduced quality of life. IBS patients often attribute their gastrointestinal effects to lactose intolerance (LI) and may avoid/limit intake of dairy products. As LI and IBS share similar symptoms, IBS patients may wrongly attribute lactose intolerance as one of the causative factors and avoid dairy products altogether. Self-imposed reductions in consumption of dairy products could reduce calcium intake leading to reduced bone mineral density. This study aims to determine the prevalence of lactose malabsorption among athletes suffering from IBS and the potential of lactose free probiotics dairy products in alleviating gastrointestinal symptoms. The inclusion of probiotics dairy products in patients' diet will be beneficial in the long term to ensure adequate intake of calcium.

DETAILED DESCRIPTION:
Irritable Bowel Syndrome (IBS) is a common, global, functional gastrointestinal disorder. It affects a significant number of people, i.e. between 9 - 23% of the world's population. The aetiology and diagnosis of IBS is poorly understood due to the complexity, heterogeneity and incomplete understanding of the pathology, thus well-defined treatments and protocols are lacking. For example, impaired motility and sensitivity, changes in gut microbiome, increased permeability, low-grade inflammation, gut endocrine cells, and alterations in the gut-brain axis, all of which are identified to play a pivotal role in the pathophysiology of IBS. Thus, it may be challenging to identify the cause of a patient's symptoms as the pathology is not fully understood. IBS can also further be divided into four subtypes based on a patient's stool patterns: constipation-predominant (IBS-C), diarrhoea-predominant (IBS-D), mixed diarrhoea and constipation (IBS-M) and those whose bowel habits cannot be identified but meet the criteria (IBS-U).

Dietary modifications in treating IBS have also received significant recognition, as many patients report that foods appear to induce or exacerbate their symptoms, thus diet intervention may be a very effective tool in the symptom management of IBS. Strategies to relief symptoms include consuming a low fermentable oligosaccharides, disaccharides, monosaccharides, and polyol (FODMAP) diet, inclusion of prebiotics and probiotics in diet. Probiotics are defined as "live microorganisms that when administered in adequate amounts, confer a health benefit to host". Previous studies suggest that consumption of probiotics help to alleviate symptoms among IBS patients. However, there is still a lack of probiotic intervention studies using lactose-free dairy products to determine the efficacy in relieving IBS symptoms. The aims of this study are (i) to determine the prevalence of lactose malabsorption among athletes suffering from IBS and (ii) to evaluate the potential of lactose free probiotics dairy products in alleviating gastrointestinal symptoms among IBS patients.

Subject recruitment Twelve to 15 recreational athletes (age > 18 years) with diagnosed irritable bowel syndrome will be recruited. A recreational athlete is defined as a person who is physically active but does not train for competition at the same level of intensity and focus as a competitive athlete. Participants will be recruited from the North West IBS support group. The study will also be opened to staff and students at the university.

Hydrogen Breath Test Participants will be asked to follow an overnight (12 hour) fasting period, not to smoke or vape for at least 24 hours prior to the test and not to exercise for at least 1 hour before taking the test. Breath testing will be conducted in Nutrition and Health Suite, Darwin Building, University of Central Lancashire to determine the baseline hydrogen breath concentration using a portable breath analyser. Participants will then be provided with 400 ml semi-skimmed milk for consumption following baseline sampling. Subsequent breath samples will then be collected for re-testing every 15 minutes for 3 hours. Lactose malabsorption is present if the peak of hydrogen breath excretion over the baseline is ≥20ppm.

Lactose-free dairy products Participants will be randomised using computer random allocation sequence into either the intervention group (lactose free probiotic yogurt) or the control group (lactose free, non-probiotic yogurt). The lactose free probiotic yogurt and lactose free non-probiotic yogurt (control) will be purchased and stored at the laboratory refrigerator the day before the testing. Only lactose free probiotic yogurt containing cultures such as Lactobacillus acidophilus and Bifidobacterium lactis will be selected. Participants will be asked to consume 125g of lactose free products daily for 7 days, followed by 1-week washout period and crossover to alternate treatment for 7 days.

Questionnaires

Participants will be asked to complete the following questionnaires at Week 0 (before the start of the dietary intervention), end of Week 1 (upon completion of 1st dietary intervention), end of Week 2 (upon completion of washout period) and end of Week 3 (upon completion of 2nd dietary intervention):

i) Participants' characteristics, records of exercise, stool frequency and consistency ii) IBS Severity Score Scale (IBS-SSS) iii) IBS Quality of Life (IBS-QOL)

ELIGIBILITY:
Inclusion Criteria:

* Recreational athlete (defined as a person who is physically active but does not train for competition at the same level of intensity and focus as a competitive athlete )
* Diagnosed with irritable bowel syndrome

Exclusion Criteria:

* Other gastrointestinal diseases such as inflammatory bowel disease, other serious chronic diseases, coeliac disease, have an allergy to product ingredients (milk), diabetic and pregnant or breastfeeding.
* unable to fast overnight, undergoing antibiotic therapies, bowel preparation for investigative procedures, and change to IBS medication during the past month prior to data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
IBS Severity Score Scale (IBS-SSS) | 3 weeks
  The IBS-SSS is a questionnaire commonly used to evaluate the severity of IBS symptoms. There are five questions (i) abdominal pain intensity; (ii) abdominal distension; (iii) bowel habit dissatisfaction, (iv) life interference and (v) abdominal pain frequency (defined as number of days with pain during the last 10 days). Higher scores indicate more severe symptoms.

SECONDARY OUTCOMES:
IBS Quality of Life (IBS-QOL) | 3 weeks
  The IBS-QOL is a questionnaire to assess the burden of IBS on participants' everyday functioning and wellbeing. The instrument consists of 34 items assessing wellbeing across eight subscales: dysphoria, activity interference, body image, social reaction, health worry, food avoidance, relationships and sexual. Respondents rate each item on a 5-point scale ranging from 1 (Not at all) to 5 (Extremely / A great deal). All items are summed to calculate the IBS-QOL total score. It is then converted to a scale of 0-100 using the following formula: [(sum of items - lowest possible score) / possible raw score range] x 100 The higher the score, the higher the health-related quality of life.
Stool frequency and consistency | 3 weeks
  Participants are provided with forms to record their stool frequency (e.g. once / twice a day) and stool consistency (e.g. Type 1, 2...7) based on Bristol stool chart.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Lancashire, Preston, United Kingdom

IPD SHARING:
Plan to Share IPD: No